CLINICAL TRIAL: NCT02832674
Title: An Open-Label, Single-Center, Single-Treatment, Safety and Effectiveness Evaluation of Percutaneous Radiofrequency in Achieving Submental Lift
Brief Title: Safety and Effectiveness Evaluation of the Device in Achieving Submental Lift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ThermiGen, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THERMI_0005
Record Dates: First submitted 2016-06-10; First posted 2016-07-14 (Estimated); Results first posted 2018-05-01 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2016-07

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Treatment (Experimental): All enrolled subjects will receive a Percutaneous Radiofrequency Single Treatment'
  Interventions: Device: Percutaneous Radiofrequency single treatment

INTERVENTIONS:
Device: Percutaneous Radiofrequency single treatment — Percutaneous Radiofrequency single treatment' under controlled temperature conditions based on pre-defined amounts of energy as controlled by the device internal algorithm, and investigator expertise. Additionally, Hunsted solution will be infused in the treatment area to eliminate the electrode/fiber to touch inner layers of the skin. External temperatures (skin surface) will be monitored using a temperature reading camera to ensure the external temperature stays within acceptable levels during the procedure Ice packs will also be used as needed to cool the treatment area based on the Thermal Camera Reading where the . heat delivery may be exceeding the threshold.
  Other Names: Thermi Percutaneous Radiofrequency Treatment; Hunsted Infusion on the treatment area; Thermal Camera; Ice packs

SUMMARY:
A prospective evaluation of the ThermiRF device in treating skin laxity under the chin and neck. Seventy male and female subjects between the age of 35 and 65 (inclusive) will be enrolled in this trial. The first 30 subjects will have a total of 6 study visits while the remainder will have a total of 5 study visits.

All subjects will have a single treatment administered. The first 30 subjects will have an extra visit at Day 60 intended to allow collection of photo images post treatment to be used for the validation of three blinded raters.

Photo images will be collected using 2D standard photography and 3D using the Vectra system. The architecture of the skin in the affected area will be measured using the Cutometer, a suction like instrument that measures elasticity. Sensory and safety will be measured using a 0-10 point numerical rating scale (NRS) and collection of safety reports. The study duration is approximately 6 months.

DETAILED DESCRIPTION:
This is an open-label, single-center, single-treatment prospective evaluation of the ThermiRF device in the treatment of submental skin laxity. The purpose of this prospective study is to determine the effectiveness and safety of the ThermiRF device in achieving overall submental lift.

In this study, "Lift" is defined as a ≥ 20 mm2 lift of the submental area after the ThermiRF treatment.

A total of 70 male and female healthy volunteers between the age of 35 and 65 will be considered for this study. Subjects who sign the informed consent form and meet all entry criteria will be enrolled in this study and will be assigned a unique number/code to preserve confidentiality.

A total of six study visits are planned as described below:

* Visit 1: Screening visit - (Day 1)
* Visit 2: Single Treatment visit
* Visit 3: Day 30 safety assessment (± 7 to 14 days)
* Visit 4: Day 60 safety and Image capture for validation exercise (± 7 to 14 days)
* Visit 5: Day 90 safety and effectiveness follow-up visit (± 7 to 14 days)
* Visit 6: Day 180 safety and effectiveness follow-up visit - (± 7 to 14 days)

Photo images (2D and 3D) will be collected at Visits 1, Visit 4 (on first 30 subjects only), and at Visits 5 and 6 using a standard camera (2D) and the Vectra system (3D). The purpose of the photos are to quantitatively and qualitative evaluate treatment effectiveness using objective and subjective assessments to measure physical changes to the skin's microstructure and aesthetic skin features over time.

A skin elasticity assessment using the Cutomer will be collected at Visits 1 (screening), 5 (Day 90) and 6 (Day 180) to assess if any biomechanical changes of the skin occurred as a result of the ThermiRF treatment.

Safety assessments will be collected using the Numerical Rating Scale (NRS) a 10-point scale, and adverse events reports (observed or reported).

The overall study duration is approximately 12 months (i.e., 5-6 month recruitment period and 6 month study visits).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the age of 35 and 65 inclusive;
* Mild to Moderate Skin Laxity Severity on the submental area defined as: "normal" muscle, "mild to moderate" skin laxity and "mild to moderate" fat;
* Desire to improve jawline definitions and/or submental skin lift
* Body mass index (BMI) ≤30;
* Females of childbearing potential who are sexually active must be willing to use an approved method of birth control during study participation.
* Cooperative, reliable, and able to read and comprehend English;
* Able to read, understand, sign and date the informed consent document (English only);
* Able and willing to comply with the schedule visit(s) and study requirements.

Exclusion Criteria:

* Excessive subcutaneous fat on the submental area
* Use within 24 hours preceding surgery of ibuprofen, acetaminophen, any other analgesics, anti-inflammatory products, or any products including herbals and supplements that could interfere with the clinical assessments of this study (other than drugs used for anesthesia);
* History of cosmetic treatments on the face and neck including but not limited to: facial skin tightening procedures within the past year, injectable fillers of any type, Botox on the lower face, ablative resurfacing laser treatment, none ablative, rejuvenative laser or light treatment within the past six months, deep facial peels, dermabrasion, face lift, neck lift, blepharoplasty or brow lift, contour threads or other.
* History or current injury to the Head and Neck.
* Severe solar elastosis
* Clinically significant facial wounds, lesions or acute infections including cystic acne, dermatitis, lupus or other immunodeficiency affecting the dermis
* Presence of metal stents or facial implants
* Pregnant or planning pregnancy prior to the end of study participation
* Current or past history of smoking
* History or current diagnosis of cancer of any type
* History of uncontrolled cardiovascular disease(i.e. myocardial infarction, hypertension, hypercholesterolemia, peripheral vascular disease, other)
* Known hypersensitivity to local anesthetic medications
* History, or current bleeding disorders (i.e. hemophilia or von Willebrand disease), or anticipated treatment with prescription anticoagulants
* Possesses a surgically implanted electronic device (i.e. pacemaker)
* History of AIDs/HIV
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to follow study subject requirement and/or record the necessary study measurements
* A family member of the investigator or an employee of the investigator.
* Participation in any other investigational study within 30 days prior to consent;

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-06-25 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry DiBernardo, MD, Principal Investigator — New Jersey Plastic Surgery; Toni Fournier, Study Director — ThermiGen, LLC; Kevin O'Brien, Study Chair — ThermiGen, LLC
Locations (1):
- New Jersey Plastic Surgery, Montclair, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred and twenty-one subjects were screened and 72 were enrolled. study initiation 25Jun2015.
Pre-assignment Details: No significant events occurred during the study recruitment process.
Period: Overall Study
Arm/Group | Single Treatment
Started | 72
Completed | 67
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Single Treatment
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 55
  More than one race | 1
  Unknown or Not Reported | 14
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.1 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Tissue Lift at the Submental Area Measuring >/= 20 mm2
Description: A >/= 20 mm^2 change from baseline at Day 90 as measured quantitatively using 3D photo images (a calculation).
Time Frame: Change from baseline at Day 90
Measure: Mean (90% Confidence Interval); unit: percentage of participants
Arm/Group | Single Treatment
Number analyzed (Participants) | 72
percentage of participants | 56.9 [46.6 to 66.9]
Statistical Analysis 1: Comparison: Single Treatment; The primary endpoint was an evaluation of the proportion of subjects with ≥ 20 mm2 lift at Day 90; Test type: Superiority; p = 0.05, Fisher Exact

2. Secondary Outcome: Percent of Participants Rated as Improved or Not Improved as Scored by the Blinded Rater/Reviewer
Description: Overall improvement of submental lift was determined by a blinded rater panel using before and after photos
Time Frame: Change from baseline to Days 90 and 180
Population: sixty-nine of the 72 enrolled and treated subjects completed visit 5 (Day 90) and 67 completed Visit 6 (Day 180). subjects with non-evaluable images were excluded from the analysis for Day 90 and 180 as applicable
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Treatment
Number analyzed (Participants) | 66
percentage of participants
  Improvement Day 90 = Yes | 74.2 [62 to 84.2]
  Improvement Day 90 = No | 25.8 [15.8 to 38]
  Improvement Day 180 = Yes: number analyzed (Participants) | 56
  Improvement Day 180 = Yes | 71.4 [57.8 to 82.7]
  Improvement Day 180 = No: number analyzed (Participants) | 56
  Improvement Day 180 = No | 28.6 [17.3 to 42.2]
Statistical Analysis 1: Comparison: Single Treatment; Test type: Other — Binomial test of proportions; p = 0.025, Chi-squared; The summary included number and percentage of subjects in each of the categories and the 2 sided Clopper-Pearson 95% CI. a binomial test of proportions tested the improvement at Day 90 and Day 180

3. Secondary Outcome: Physician Global Aesthetic Improvement Scale (P-GAIS)
Description: A subjective assessment of overall improvement measured by the physician using the PGAIS where the physician rates the appearance of the treated area (submental area) with respect to lift compared to baseline photography at the defined time points. The 5-point scale measures from "Very much improved" to "worse".
Time Frame: Change from baseline at Days 90 and 180
Population: of the 72 enrolled and treated subjects, 69 completed Day 90 and 67 completed the Day 180 visit (4 subjects were lost to follow up and 1 withdrew consent)
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Treatment
Number analyzed (Participants) | 69
percentage of participants
  Improvement Day 90 = Yes | 94.2 [85.8 to 98.4]
  Improvement Day 90 = No | 5.8 [1.6 to 14.2]
  Improvement Day 180 = Yes: number analyzed (Participants) | 67
  Improvement Day 180 = Yes | 89.6 [79.7 to 95.7]
  Improvement Day 180 = No: number analyzed (Participants) | 67
  Improvement Day 180 = No | 10.4 [4.3 to 20.3]
Statistical Analysis 1: Comparison: Single Treatment; Analysis of all effectiveness endpoints was conducted on the ITT population and on the PP population; Test type: Other; p = 0.025, Chi-squared; [other analysis details as in outcome 2, analysis 1]

4. Secondary Outcome: Subject Global Aesthetic Improvement Scale (S-GAIS)
Description: A subjective assessment of overall improvement measured by the participant using the SGAIS where the participant rates the appearance of the treated area (submental area) with respect to "lift"is measured from. the 5-point scale measures from Very much improved to worse.
Time Frame: Change from baseline at Days 90 and 180
Population: of the 72 enrolled and treated subjects, 69 completed the Day 90 visit and 67 completed day 180 (4 subjects were lost to follow up and 1 subject withdrew consent)
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Treatment
Number analyzed (Participants) | 69
percentage of participants
  Improvement Day 90 = Yes | 89.9 [80.2 to 95.8]
  Improvement Day 90 = No | 10.1 [4.2 to 19.8]
  Improvement Day 180 = Yes: number analyzed (Participants) | 67
  Improvement Day 180 = Yes | 83.6 [72.5 to 91.5]
  Improvement Day 180 = No: number analyzed (Participants) | 67
  Improvement Day 180 = No | 16.4 [8.5 to 27.5]
Statistical Analysis 1: Comparison: Single Treatment; Test type: Other; p = 0.025, Chi-squared; [other analysis details as in outcome 2, analysis 1]

5. Secondary Outcome: Physician Global Satisfaction Questionnaire (P-GSQ)
Description: A subjective assessment of global satisfaction as measured by the physician using the P-GSQ where the physician rates his/her level of satisfaction of the treatment and treated area based on 4 satisfaction questions respective to 1. changes to the treated area, 2. skin texture of the treated area, 3. satisfaction with treatment results and 4. likelihood to recommend the treatment as a treatment option.
Time Frame: Change from baseline at Days 90 and 180
Population: Of the 72 enrolled and treated subjects, 69 completed the Day 90 visit and 67 the Day 180 (4 subjects were lost to follow up and one withdrew consent).
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Treatment
Number analyzed (Participants) | 69
percentage of participants
  Improvement Day 90 = Yes | 92.8 [83.9 to 97.6]
  Improvement Day 90 = No | 7.2 [2.4 to 16.1]
  Improvement Day 180 = Yes: number analyzed (Participants) | 67
  Improvement Day 180 = Yes | 91 [81.5 to 96.6]
  Improvement Day 180 = No: number analyzed (Participants) | 67
  Improvement Day 180 = No | 9 [3.4 to 18.5]
  Satisfaction Day 90 = Yes | 81.2 [69.9 to 89.6]
  Satisfaction Day 90 = No | 18.8 [10.4 to 30.1]
  Satisfaction Day 180 = Yes: number analyzed (Participants) | 67
  Satisfaction Day 180 = Yes | 71.6 [59.3 to 82]
  Satisfaction Day 180 = No: number analyzed (Participants) | 67
  Satisfaction Day 180 = No | 28.4 [18 to 40.7]
Statistical Analysis 1: Comparison: Single Treatment; Test type: Other; p = 0.025, Chi-squared; [other analysis details as in outcome 2, analysis 1]

6. Secondary Outcome: Subject Global Satisfaction Questionnaire (S-GSQ)
Description: A subjective assessment of global satisfaction as measured by the participant using the S-GSQ where the participant rates his/her level of satisfaction of the treatment and treated area based on 4 satisfaction questions respective to 1. changes to the treated area, 2. skin texture of the treated area, 3. satisfaction with treatment results and 4. likelihood to recommend the treatment as a treatment option.
Time Frame: Change from baseline at Days 90 and 180
Population: Of the 72 enrolled and treated subjects, 69 completed the day 90 visit and 67 completed the day 180 visit (4 subjects were lost to follow up and one subject withdrew consent)
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Single Treatment
Number analyzed (Participants) | 69
percentage of participants
  Improvement Day 90 = Yes | 88.4 [78.4 to 94.9]
  Improvement Day 90 = No | 11.6 [5.1 to 21.6]
  Improvement Day 180 = Yes: number analyzed (Participants) | 67
  Improvement Day 180 = Yes | 83.6 [72.5 to 91.5]
  Improvement Day 180 = No: number analyzed (Participants) | 67
  Improvement Day 180 = No | 16.4 [8.5 to 27.5]
  Satisfaction Day 90 = Yes | 68.1 [55.8 to 78.8]
  Satisfaction Day 90 = No | 31.9 [21.2 to 44.1]
  Satisfaction Day 180 = Yes: number analyzed (Participants) | 67
  Satisfaction Day 180 = Yes | 65.7 [53.1 to 76.8]
  Satisfaction Day 180 = No: number analyzed (Participants) | 67
  Satisfaction Day 180 = No | 34.3 [23.2 to 46.9]
Statistical Analysis 1: Comparison: Single Treatment; Test type: Other; p = 0.025, Chi-squared; [other analysis details as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time the subject signed the informed consent to last subject last visit. Duration was approximately 1.25 years.
Arm/Group | Single Treatment
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 1/72
Other Adverse Events (participants affected / at risk) | 32/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Treatment (N=72)
Retropharyngeal Swelling/Fluid (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Subject presented to the emergency room on Day 4th post treatment with pain. subject was admitted to the hospital for an unknown number of days. The event resolved two days later and the subject remained in the study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Treatment (N=72)
Application Site Hypoaesthesia (General disorders) | 22 (23)
Application Site Edema (General disorders) | 16 (17)
Application Site Pain (Gastrointestinal disorders) | 7 (7)
Application Site Swelling (General disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-05-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT02832674/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT02832674/SAP_001.pdf